CLINICAL TRIAL: NCT07096219
Title: The Improvement Effect of Catheter Ablation on Functional Mitral Regurgitation in Patients With Persistent Atrial Fibrillation and the Construction and Validation of a Predictive Model: A Multicenter Prospective Cohort Study
Brief Title: Catheter Ablation for Functional Mitral Regurgitation in Persistent Atrial Fibrillation: Development and Validation of a Predictive Model-A Multicenter Prospective Cohort Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Shantou Central Hospital (Other); Dongguan People's Hospital (Other Government); Second Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Shantou University Medical College (Other); West China Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); Qingyuan People's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Jiangmen Central Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Jiangxi Provincial People's Hopital (Other); Guangdong Provincial People's Hospital (Other); Nanhai District People's Hospital of Foshan City (Unknown); The University of Hong Kong-Shenzhen Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Second Xiangya Hospital of Central South University (Other); Zhongnan Hospital (Other); Ningbo Medical Center Li Huili Hospital (Unknown); Sir Run Run Shaw Hospital (Other); China-Japan Union Hospital, Jilin University (Other); Xiangya Hospital of Central South University (Other); Shanxi Cardiovascular Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Shenzhen People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Tongji Hospital (Other); Nanfang Hospital, Southern Medical University (Other); First People's Hospital of Foshan (Other); Renmin Hospital of Wuhan University (Other); Guizhou Provincial People's Hospital (Other); The First Affiliated Hospital of Air Force Medical University (Unknown); The First Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Jiangsu Provincial People's Hospital (Other); Meizhou People's Hospital (Other); Yuebei People's Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yangxin Chen, Chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-803-02; SYSKY-2024-803-01 (Other: SunYatsenU2H)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: AF Ablation Patients With Moderate+ FMR and Persistent AF
MeSH Terms: interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Catheter Ablation for Functional Mitral Regurgitation in Persistent Atrial Fibrillation
  Interventions: Procedure: Catheter Ablation; Diagnostic Test: ultrasonic cardiography (UCG)

INTERVENTIONS:
Procedure: Catheter Ablation — A minimally invasive procedure that delivers energy through catheters to destroy abnormal cardiac tissue causing arrhythmias.
Diagnostic Test: ultrasonic cardiography (UCG) — Trans-thoracic echocardiography (TTE) is performed in the resting position. Trans-esophageal echocardiography (TEE) is performed under surfa

SUMMARY:
Mitral Regurgitation (MR) is the most prevalent type of valvular heart disease in clinical practice, with an average prevalence of approximately 1% in populations with moderate-to-severe or worse MR, which increases significantly with age. Functional MR (FMR) is one subtype of MR and can be further classified into atrial FMR, ventricular FMR, and mixed FMR based on its underlying mechanisms. Pathophysiologically, FMR is closely associated with atrial fibrillation (AF) and heart failure (HF). Studies suggest that catheter ablation for AF may improve FMR in some patients and reverse left atrial (LA) and left ventricular (LV) remodeling. However, there is currently a lack of precise and effective indicators or predictive models to determine the evolution of FMR after AF ablation in both domestic and international research.

This study aims to conduct a multicenter prospective cohort study, enrolling patients with moderate or worse FMR and persistent AF undergoing ablation. Using postoperative 3-month FMR improvement as the primary outcome, we will employ big data mining and multimodal analysis to construct a predictive model for FMR progression after AF ablation and validate it through prospective multicenter testing. The findings will provide a scientific basis for clinical decision-making and precision medicine in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years
2. Diagnosis of functional mitral regurgitation (FMR) by transthoracic echocardiography (TTE) and/or transesophageal echocardiography (TEE) with combined qualitative and quantitative assessment, demonstrating moderate or worse regurgitation (≥ grade 2+)
3. Persistent atrial fibrillation (AF) with successful catheter ablation
4. Signed informed consent with commitment to regular follow-up for ≥1 year

Exclusion Criteria:

1. Acute or chronic degenerative mitral regurgitation (DMR) from any etiology
2. Paroxysmal or permanent atrial fibrillation
3. Planned repeat ablation for AF recurrence
4. Concomitant moderate/severe valvular disease (e.g., mitral stenosis, aortic stenosis/regurgitation, pulmonary stenosis/regurgitation)
5. Prior valvular surgery/intervention
6. History of open-heart surgery
7. Severe pulmonary hypertension (PASP >70 mmHg) refractory to medical therapy
8. Left atrial diameter ≥60 mm (diastolic phase) on echocardiography
9. Uncontrolled hyperthyroidism
10. Intracardiac mass/thrombus/vegetation
11. Significant shunts (ASD/VSD/PDA)
12. Hypertrophic obstructive cardiomyopathy
13. Active severe infection/sepsis (including infective endocarditis)
14. Scheduled CRT/CRT-D/CCM implantation
15. Untreated critical CAD (e.g., ≥70% stenosis in proximal/mid LAD/LCX/RCA requiring revascularization) or concomitant major cardiovascular surgery needs
16. End-stage heart failure (ACC/AHA Stage D) requiring mechanical support/transplant listing
17. Severe hepatic dysfunction (acute liver failure/decompensated cirrhosis, Child-Pugh C)
18. Severe renal impairment (CKD 5: eGFR<15 mL/min or dialysis)
19. Hemodynamic instability (SBP<90 mmHg/MAP<70 mmHg with hypoperfusion [urine output<30 mL/h])
20. Contraindications to antithrombotics: Active bleeding (GI/intracranial/visceral), bleeding disorders (hemophilia/ITP/leukemia etc.), severe hematologic abnormalities (platelets<20×10⁹/L, spontaneous INR>3)
21. Uncontrolled autoimmune/connective tissue disease
22. Acute MI within 4 weeks
23. Stroke within 30 days
24. Acute peptic ulcer/upper GI bleeding within 3 months
25. Pregnancy/lactation
26. Declined informed consent
27. Life expectancy <1 year
28. Poor compliance (anticipated inability to complete follow-up)
29. Concurrent participation in conflicting clinical trials
30. Other investigator-determined exclusions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate-to-severe functional mitral regurgitation (FMR) and persistent atrial fibrillation undergoing catheter ablation
Sampling Method: Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was MR improvement at 3 months post-procedure. | From the operation day to 3 months after operation.
  MR improvement was defined as a reduction in regurgitation severity by ≥1 grade on 3-month post-ablation transthoracic echocardiography (TTE) compared to baseline. Absence of improvement or worsening was categorized as non-improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Yangxin Chen, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No